CLINICAL TRIAL: NCT02693392
Title: Clinical Evaluation of Fenugreek Seed Extract, a Nutraceutical in Patients With Type- 2 Diabetes: An Add-On Study
Brief Title: Clinical Evaluation of Fenugreek Seed Extract, a Nutraceutical in Patients With Type- 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Collaborators: Chemical Resources (Industry)
Responsible Party: Principal Investigator, Dr Debasish Hota, Professor & Head, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: T/EM-F/Pharma/14/05
Record Dates: First submitted 2016-02-19; First posted 2016-02-26 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Type-2 Diabetes Mellitus
Keywords: Fenugreek seed extract; HbA1c; Blood glucose
MeSH Terms: interventions — Hypoglycemic Agents; Metformin; Sulfonylurea Compounds; fenugreek seed meal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): One hundred type-2 diabetes patients with standard oral hypoglycemic drugs (metformin +/- sulfonylurea) will be recruited and followed up without add-on fenugreek extract.
  Interventions: Drug: Oral hypoglycemic agents (pre-specified) [Metformin, Sulfonylurea]
- Fenugreek (Experimental): One hundred type-2 diabetes patients with standard oral hypoglycemic drugs (metformin +/- sulfonylurea) will be recruited and followed up with add-on fenugreek extract.
  Interventions: Drug: Oral hypoglycemic agents (pre-specified) [Metformin, Sulfonylurea]; Dietary Supplement: Fenugreek Seed extract

INTERVENTIONS:
Drug: Oral hypoglycemic agents (pre-specified) [Metformin, Sulfonylurea] — Patients receiving either of the following oral hypoglycemic agents
  1. Sulfonylurea based oral hypoglycemic agents
  2. Metformin based oral hypoglycemic agents
  3. Metformin plus Sulfonylurea based oral hypoglycemic agents
  Other Names: Metformin, Sulfonylurea
Dietary Supplement: Fenugreek Seed extract — Patients recruited in the study arm will receive Capsule Fenfuro 500 milligram twice daily for 12 weeks as add-on intervention to the pre-specified oral hypoglycemic agents therapy
  Other Names: Capsule Fenfuro 500 mg
  Arms: Fenugreek

SUMMARY:
In the proposed study, hydroalcoholic Fenugreek seed extract will used add-on to the existing therapy in patients with type-2 diabetes. The efficacy and safety of the extract will be evaluated using standard methodology.

DETAILED DESCRIPTION:
Trigonella foenum-graecum, commonly known as Fenugreek, is a plant that has been extensively used as a source of antidiabetic compounds, from its seeds, leaves and extracts in different systems of medicine in asia. Fenugreek is traditionally used in India, especially in the Ayurvedic and Unani systems. Preliminary animal and human studies suggest possible hypoglycemic and anti-hyperlipidemic properties of fenugreek seed powder taken orally. In a randomized placebo controlled study conducted by Gupta et al showed that two month treatment with the hydro-alcoholic extract of fenugreek seeds improved glycemic control in 12 non-insulin dependent diabetes mellitus patients. In addition, there was improvement in insulin sensitivity and plasma lipid profile. Fenugreek extract was also well tolerated in diabetic patients.

In the proposed study, hydroalcoholic Fenugreek seed extract will used add-on to the existing therapy in patients with type-2 diabetes. The efficacy and safety of the extract will be evaluated using standard methodology.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Type-2 Diabetes of less than 10 years duration
* Patients with HbA1c >7.0%
* Patients with fasting plasma glucose not exceeding 180 mg/dL
* Patients with Negative Urine sugar
* Patients who are on oral hypoglycaemic agents containing either Metformin or Sulfonylurea or both
* There should not be any change their in anti-diabetic treatment for at least one month

Exclusion Criteria:

* Patients with diabetes other than type-2 diabetes mellitus
* Patients with evidence of renal disease (S. Creatinine > 1.5mg/dL)
* Patients with evidence of liver disease (AST/ALT >3 times of normal
* Pregnant and lactating mothers and women intending pregnancy
* Patients who participated in any other clinical trial within the last 30 days
* Patients with history of any hemoglobinopathy
* History of intolerance or hypersensitivity to Fenugreek

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-01-17 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-08-16 (Actual)

PRIMARY OUTCOMES:
Glycosylated hemoglobin (HbA1c) | Change from baseline HbA1c over 12 weeks
  HbA1c will be evaluated using Hb variant (HPLC)

SECONDARY OUTCOMES:
Fasting blood glucose | Change from baseline Fasting Blood Glucose over 12 weeks
  METHOD : SPECTROPHOTOMETRY HEXOKINASE
Serum Insulin | Change from baseline Serum Insulin over 12 weeks
  by CHEMILUMINESCENCE method
Serum C-Peptide | Change from baseline Serum C-Peptide over 12 weeks
  by CHEMILUMINESCENCE method
Renal Function Test | Change from baseline Renal function test over 12 weeks
  by Spectrophotometry
Liver Function Test | Change from baseline Liver function test over 12 weeks
  by Spectrophotometry
Hematology (whole blood cell count) | Change from baseline Hematology over 12 weeks
  Automated particle cell counter and microscopy
Urinary sugar | Change from baseline Urinary over 12 weeks
  Semi-quantitative Biochemical test
Post-prandial Blood Glucose | Change from baseline post-prandial Blood Glucose over 12 weeks
  METHOD: SPECTROPHOTOMETRY HEXOKINASE

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine and Department of Pharmacology, AIIMS, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gupta A, Gupta R, Lal B. Effect of Trigonella foenum-graecum (fenugreek) seeds on glycaemic control and insulin resistance in type 2 diabetes mellitus: a double blind placebo controlled study. J Assoc Physicians India. 2001 Nov;49:1057-61. PMID 11868855
- [Result] Neelakantan N, Narayanan M, de Souza RJ, van Dam RM. Effect of fenugreek (Trigonella foenum-graecum L.) intake on glycemia: a meta-analysis of clinical trials. Nutr J. 2014 Jan 18;13:7. doi: 10.1186/1475-2891-13-7. PMID 24438170
- [Result] Baquer NZ, Kumar P, Taha A, Kale RK, Cowsik SM, McLean P. Metabolic and molecular action of Trigonella foenum-graecum (fenugreek) and trace metals in experimental diabetic tissues. J Biosci. 2011 Jun;36(2):383-96. doi: 10.1007/s12038-011-9042-0. PMID 21654091
- [Result] Hannan JM, Ali L, Rokeya B, Khaleque J, Akhter M, Flatt PR, Abdel-Wahab YH. Soluble dietary fibre fraction of Trigonella foenum-graecum (fenugreek) seed improves glucose homeostasis in animal models of type 1 and type 2 diabetes by delaying carbohydrate digestion and absorption, and enhancing insulin action. Br J Nutr. 2007 Mar;97(3):514-21. doi: 10.1017/S0007114507657869. PMID 17313713